CLINICAL TRIAL: NCT00446043
Title: A Long-term Safety and Efficacy Study of a Fixed Combination of Adapalene 0.1% and Benzoyl Peroxide 2.5% (Adapalene and Benzoyl Peroxide Topical Gel) Gel in Subjects With Acne Vulgaris
Brief Title: Long-term Study of Efficacy/Safety of Adapalene/Benzoyl Peroxide Topical Gel in Acne Vulgaris Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RD.06.SPR.18089
Record Dates: First submitted 2007-03-08; First posted 2007-03-12 (Estimated); Results first posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2022-08

CONDITIONS: Acne Vulgaris
Keywords: Acne Vulgaris; Adapalene; Benzoyl Peroxide
MeSH Terms: conditions — Acne Vulgaris | interventions — Adapalene, Benzoyl Peroxide Drug Combination

ARMS (1):
- Adapalene/Benzoyl Peroxide (Experimental): Participants were treated with adapalene 0.1 percent (%) [weight by weight (W/W)] and benzoyl peroxide 2.5 percent (%) (W/W) gel topically to the face and trunk area once daily in the evening.
  Interventions: Drug: Adapalene/Benzoyl Peroxide

INTERVENTIONS:
Drug: Adapalene/Benzoyl Peroxide — Adapalene 0.1 percent (%) [weight by weight (W/W)] and benzoyl peroxide 2.5 % (W/W) gel topically daily in the evening.

SUMMARY:
This was a multi-center, open-label, non-comparative study that evaluated the long-term safety and efficacy profile of Adapalene/Benzoyl Peroxide Gel.

Subjects were evaluated at Baseline, Weeks 1 and 2, and Months 1, 2, 4, 6, 8, 10, and 12.

Safety was evaluated by spontaneous reports of Adverse Events (AEs), the Local Tolerability Assessment (Erythema, Scaling, Dryness, and Stinging/Burning), routine laboratory testing (hematology, blood chemistry, and urinalysis), and monitoring of suspected sensitizations. Efficacy was evaluated by analysis of Percent Change from Baseline in Inflammatory, Noninflammatory, and Total Lesion Counts, and by the Subject's Assessment of Acne.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of acne vulgaris with facial involvement.
* A minimum of 20 but not more than 50 Inflammatory lesions.
* A minimum of 30 but not more than 100 Noninflammatory lesions.

Exclusion Criteria:

* Subjects with presence of nodules or cysts.
* Acne conglobate, acne fulminans, secondary acne, or severe acne.
* Underlying diseases that required the use of interfering topical or systemic therapy.
* Use of prohibited medications prior to the study unless appropriate washout period was documented.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 452 (Actual)
Dates: Start 2004-02-17 (Actual); Primary Completion 2005-05-23 (Actual); Study Completion 2005-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Graeber, MD, Study Director — Galderma R&D
Locations (1):
- Phoebe Rich, MD, Portland, Oregon, United States

REFERENCES:
- [Background] Leyden JJ. A review of the use of combination therapies for the treatment of acne vulgaris. J Am Acad Dermatol. 2003 Sep;49(3 Suppl):S200-10. doi: 10.1067/s0190-9622(03)01154-x. PMID 12963896

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 452 participants were enrolled at 28 study centers in the United States from 17 February 2004 to 23 May 2005.
Groups:
- Adapalene/Benzoyl Peroxide: Participants were treated with adapalene 0.1 percent (%) [weight by weight (W/W)] and benzoyl peroxide 2.5% (W/W) gel topically to the face and trunk area as applicable once daily in the evening.
Period: Overall Study
Arm/Group | Adapalene/Benzoyl Peroxide
Started | 452
Completed | 327
Not Completed | 125
Not completed — Adverse Event | 9
Not completed — Withdrawal by Subject | 70
Not completed — Protocol Violation | 2
Not completed — Lost to Follow-up | 42
Not completed — Pregnancy | 2

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population included all participants who were enrolled and to whom medication was dispensed.
Groups:
- Adapalene/Benzoyl Peroxide: Participants were treated with adapalene 0.1 % (W/W) and benzoyl peroxide 2.5 % (W/W) gel topically to the face and trunk area as applicable once daily in the evening.
Arm/Group | Adapalene/Benzoyl Peroxide
Number analyzed (Participants) | 452
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.3 (6.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 230
  Male | 222
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian | 345
  Race: Black | 53
  Race: Asian | 10
  Race: Hispanic | 31
  Race: Other | 13

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Inflammatory, Noninflammatory and Total Lesion Count at Month 12 LOCF
Description: Percent change in inflammatory, noninflammatory and total lesions at Month 12 was measured from baseline lesions. The noninflammatory lesion count was the sum of open comedones (a mass of sebaceous material that is impacted behind an open follicular orifice (blackhead) and closed comedones (a mass of sebaceous material that is impacted behind a closed follicular orifice (whitehead). The inflammatory lesion count was the sum of papules (a small, solid elevation less than 1.0 cm in diameter) and pustules (a small, circumscribed elevation of the skin that contains yellow-white exudate). The total lesion count was the sum of inflammatory and noninflammatory lesions. Missing adapalene and benzoyl peroxide data were imputed using last observation carried forward (LOCF).
Time Frame: Baseline, Month 12 LOCF
Population: ITT population included all participants who were enrolled and treated to whom medication was dispensed.
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Adapalene/Benzoyl Peroxide: Participants were treated with adapalene 0.1% (W/W) and benzoyl peroxide 2.5 % (W/W) gel topically to the face and trunk area, as applicable, once daily in the evening.
Arm/Group | Adapalene/Benzoyl Peroxide
Number analyzed (Participants) | 452
percent change
  Inflammatory Lesion Counts | -59.70 (34.268)
  Noninflammatory Lesion Counts | -58.80 (33.206)
  Total Lesion Counts | -58.85 (29.273)

2. Primary Outcome: Number of Participants Categorized Based on Participant's Assessment Scale of Acne at Month 6
Description: Participant's assessment of acne improvement was graded as 0; complete improvement, 1; marked improvement, 2; moderate improvement, 3; minimal improvement, 4; no change, 5; worse.
Time Frame: At Month 6
Population: ITT population included all participants who were enrolled and to whom medication was dispensed. Here, "overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- Adapalene/Benzoyl Peroxide: Participants were treated with adapalene 0.1 % (W/W) and benzoyl peroxide 2.5 % (W/W) gel topically to the face and trunk area, as applicable, once daily in the evening.
Arm/Group | Adapalene/Benzoyl Peroxide
Number analyzed (Participants) | 359
Participants
  0=Complete Improvement | 17
  1=Marked Improvement | 149
  2=Moderate Improvement | 147
  3=Minimal Improvement | 31
  4=No Change | 11
  5=Worse | 4

3. Primary Outcome: Number of Participants Categorized Based on Participant's Assessment Scale of Acne at Month 12
Description: as for outcome 2
Time Frame: At Month 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Adapalene/Benzoyl Peroxide
Number analyzed (Participants) | 327
Participants
  0=Complete Improvement | 40
  1=Marked Improvement | 164
  2=Moderate Improvement | 77
  3=Minimal Improvement | 37
  4=No Change | 6
  5=Worse | 3

4. Secondary Outcome: Number of Participants With Local Tolerability Assessment For Erythema
Description: Local tolerability assessment for erythema (abnormal redness of the skin) was graded on a "0" (none) to "3" (severe) scale as follows; none (0- no erythema), mild (1- slight pinkness present), moderate (2- definite redness, easily recognized), severe (3- intense redness). The worst severity scores were generally mild or moderate, and rarely severe.
Time Frame: Baseline, Weeks 1 and 2, Months 1, 2, 4, 6, 8, 10 and 12
Population: The safety population was defined as all participants enrolled who had applied study medication at least once. Here, 'number analyzed' signifies participants who were evaluable at each post-baseline timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Adapalene/Benzoyl Peroxide
Number analyzed (Participants) | 452
Participants
  Baseline: 0 = None | 348
  Baseline: 1 = Mild | 94
  Baseline: 2=Moderate | 10
  Baseline: 3=Severe | 0
  Week 1: number analyzed (Participants) | 423
  Week 1: 0 = None | 233
  Week 1: 1 = Mild | 157
  Week 1: 2=Moderate | 32
  Week 1: 3=Severe | 1
  Week 2: number analyzed (Participants) | 429
  Week 2: 0 = None | 277
  Week 2: 1 = Mild | 133
  Week 2: 2=Moderate | 17
  Week 2: 3=Severe | 2
  Month 1: number analyzed (Participants) | 415
  Month 1: 0 = None | 292
  Month 1: 1 = Mild | 105
  Month 1: 2=Moderate | 18
  Month 1: 3=Severe | 0
  Month 2: number analyzed (Participants) | 426
  Month 2: 0 = None | 320
  Month 2: 1 = Mild | 90
  Month 2: 2=Moderate | 16
  Month 2: 3=Severe | 0
  Month 4: number analyzed (Participants) | 389
  Month 4: 0 = None | 334
  Month 4: 1 = Mild | 48
  Month 4: 2=Moderate | 7
  Month 4: 3=Severe | 0
  Month 6: number analyzed (Participants) | 361
  Month 6: 0 = None | 296
  Month 6: 1 = Mild | 59
  Month 6: 2=Moderate | 6
  Month 6: 3=Severe | 0
  Month 8: number analyzed (Participants) | 341
  Month 8: 0 = None | 276
  Month 8: 1 = Mild | 57
  Month 8: 2=Moderate | 8
  Month 8: 3=Severe | 0
  Month 10: number analyzed (Participants) | 329
  Month 10: 0 = None | 270
  Month 10: 1 = Mild | 56
  Month 10: 2=Moderate | 3
  Month 10: 3=Severe | 0
  Month 12: number analyzed (Participants) | 327
  Month 12: 0 = None | 284
  Month 12: 1 = Mild | 39
  Month 12: 2=Moderate | 4
  Month 12: 3=Severe | 0

5. Secondary Outcome: Number of Participants With Local Tolerability Assessment For Scaling
Description: Local tolerability assessment for scaling (abnormal shedding of the stratum corneum) was graded on a "0" (none) to "3" (severe) scale as follow; none (0- no Scaling), mild (1- barely perceptible shedding, noticeable only on light scratching or rubbing), moderate (2- obvious but not profuse shedding), severe (3- heavy scale production).
Time Frame: Baseline, Weeks 1 and 2, Months 1, 2, 4, 6, 8, 10 and 12
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Adapalene/Benzoyl Peroxide
Number analyzed (Participants) | 452
Participants
  Baseline: 0=None | 410
  Baseline: 1=Mild | 41
  Baseline: 2=Moderate | 1
  Baseline: 3=Severe | 0
  Week 1: number analyzed (Participants) | 423
  Week 1: 0=None | 228
  Week 1: 1=Mild | 164
  Week 1: 2=Moderate | 30
  Week 1: 3=Severe | 1
  Week 2: number analyzed (Participants) | 429
  Week 2: 0=None | 284
  Week 2: 1=Mild | 130
  Week 2: 2=Moderate | 14
  Week 2: 3=Severe | 1
  Month 1: number analyzed (Participants) | 415
  Month 1: 0=None | 312
  Month 1: 1=Mild | 93
  Month 1: 2=Moderate | 10
  Month 1: 3=Severe | 0
  Month 2: number analyzed (Participants) | 426
  Month 2: 0=None | 338
  Month 2: 1=Mild | 84
  Month 2: 2=Moderate | 4
  Month 2: 3=Severe | 0
  Month 4: number analyzed (Participants) | 389
  Month 4: 0=None | 351
  Month 4: 1=Mild | 38
  Month 4: 2=Moderate | 0
  Month 4: 3=Severe | 0
  Month 6: number analyzed (Participants) | 361
  Month 6: 0=None | 330
  Month 6: 1=Mild | 28
  Month 6: 2=Moderate | 3
  Month 6: 3=Severe | 0
  Month 8: number analyzed (Participants) | 341
  Month 8: 0=None | 301
  Month 8: 1=Mild | 38
  Month 8: 2=Moderate | 2
  Month 8: 3=Severe | 0
  Month 10: number analyzed (Participants) | 329
  Month 10: 0=None | 294
  Month 10: 1=Mild | 33
  Month 10: 2=Moderate | 2
  Month 10: 3=Severe | 0
  Month 12: number analyzed (Participants) | 327
  Month 12: 0=None | 308
  Month 12: 1=Mild | 19
  Month 12: 2=Moderate | 0
  Month 12: 3=Severe | 0

6. Secondary Outcome: Number of Participants With Local Tolerability Assessment For Dryness
Description: Local tolerability assessment for dryness (brittle and/or tight sensation) was graded on a "0" (none) to "3" (severe) scale as follows; none (0- no dryness), mild (1- slight but definite roughness), moderate (2 -moderate roughness), severe (3- marked roughness).
Time Frame: Baseline, Weeks 1 and 2, Months 1, 2, 4, 6, 8, 10 and 12
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Adapalene/Benzoyl Peroxide
Number analyzed (Participants) | 452
Participants
  Baseline: 0=None | 385
  Baseline: 1=Mild | 65
  Baseline: 2=Moderate | 2
  Baseline: 3=Severe | 0
  Week 1: number analyzed (Participants) | 423
  Week 1: 0=None | 195
  Week 1: 1=Mild | 190
  Week 1: 2=Moderate | 35
  Week 1: 3=Severe | 3
  Week 2: number analyzed (Participants) | 429
  Week 2: 0=None | 264
  Week 2: 1=Mild | 152
  Week 2: 2=Moderate | 12
  Week 2: 3=Severe | 1
  Month 1: number analyzed (Participants) | 415
  Month 1: 0=None | 281
  Month 1: 1=Mild | 121
  Month 1: 2=Moderate | 12
  Month 1: 3=Severe | 1
  Month 2: number analyzed (Participants) | 426
  Month 2: 0=None | 311
  Month 2: 1=Mild | 109
  Month 2: 2=Moderate | 6
  Month 2: 3=Severe | 0
  Month 4: number analyzed (Participants) | 389
  Month 4: 0=None | 337
  Month 4: 1=Mild | 52
  Month 4: 2=Moderate | 0
  Month 4: 3=Severe | 0
  Month 6: number analyzed (Participants) | 361
  Month 6: 0=None | 320
  Month 6: 1=Mild | 37
  Month 6: 2=Moderate | 4
  Month 6: 3=Severe | 0
  Month 8: number analyzed (Participants) | 341
  Month 8: 0=None | 281
  Month 8: 1=Mild | 58
  Month 8: 2=Moderate | 2
  Month 8: 3=Severe | 0
  Month 10: number analyzed (Participants) | 329
  Month 10: 0=None | 278
  Month 10: 1=Mild | 48
  Month 10: 2=Moderate | 3
  Month 10: 3=Severe | 0
  Month 12: number analyzed (Participants) | 327
  Month 12: 0=None | 291
  Month 12: 1=Mild | 36
  Month 12: 2=Moderate | 0
  Month 12: 3=Severe | 0

7. Secondary Outcome: Number of Participants With Local Tolerability Assessment For Stinging/Burning
Description: Local tolerability assessment for stinging/burning [prickling pain sensation immediately after (within 5 minutes of) dosing] was graded on a "0" (none) to "3" (severe) scale as follows; none (0- no stinging/ burning), mild (1- slight warm, tingling/stinging sensation; not really bothersome), moderate (2- definite warm, tingling/stinging sensation that is somewhat), severe (3- hot, tingling/stinging sensation that has caused definite discomfort).
Time Frame: Baseline, Weeks 1 and 2, Months 1, 2, 4, 6, 8, 10 and 12
Population: ITT safety population was defined as all participants enrolled who had applied study medication at least once. Here, 'number analyzed' signifies participants who were evaluable at each post-baseline timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Adapalene/Benzoyl Peroxide
Number analyzed (Participants) | 452
Participants
  Baseline: 0=None | 440
  Baseline: 1=Mild | 10
  Baseline: 2=Moderate | 2
  Baseline: 3=Severe | 0
  Week 1: number analyzed (Participants) | 423
  Week 1: 0=None | 201
  Week 1: 1=Mild | 154
  Week 1: 2=Moderate | 63
  Week 1: 3=Severe | 5
  Week 2: number analyzed (Participants) | 429
  Week 2: 0=None | 319
  Week 2: 1=Mild | 84
  Week 2: 2=Moderate | 21
  Week 2: 3=Severe | 5
  Month 1: number analyzed (Participants) | 415
  Month 1: 0=None | 331
  Month 1: 1=Mild | 66
  Month 1: 2=Moderate | 14
  Month 1: 3=Severe | 4
  Month 2: number analyzed (Participants) | 426
  Month 2: 0=None | 373
  Month 2: 1=Mild | 42
  Month 2: 2=Moderate | 10
  Month 2: 3=Severe | 1
  Month 4: number analyzed (Participants) | 389
  Month 4: 0=None | 364
  Month 4: 1=Mild | 23
  Month 4: 2=Moderate | 2
  Month 4: 3=Severe | 0
  Month 6: number analyzed (Participants) | 361
  Month 6: 0=None | 337
  Month 6: 1=Mild | 20
  Month 6: 2=Moderate | 4
  Month 6: 3=Severe | 0
  Month 8: number analyzed (Participants) | 341
  Month 8: 0=None | 312
  Month 8: 1=Mild | 23
  Month 8: 2=Moderate | 5
  Month 8: 3=Severe | 1
  Month 10: number analyzed (Participants) | 329
  Month 10: 0=None | 303
  Month 10: 1=Mild | 22
  Month 10: 2=Moderate | 4
  Month 10: 3=Severe | 0
  Month 12: number analyzed (Participants) | 327
  Month 12: 0=None | 306
  Month 12: 1=Mild | 19
  Month 12: 2=Moderate | 1
  Month 12: 3=Severe | 1

8. Secondary Outcome: Number of Participant With Adverse Event (AE) and Serious Adverse Event (SAE)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Baseline up to Month 14
Population: The safety population was defined as all participants enrolled who had applied study medication at least once.
Measure: Count of Participants; unit: Participants
Arm/Group | Adapalene/Benzoyl Peroxide
Number analyzed (Participants) | 452
Participants
  Participants (N) With At least one AE | 288
  Participants (N) With At Least one SAE | 5

9. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Laboratory Parameters
Description: Clinical laboratory parameters included hematology, blood chemistry, urinalysis. Number of participants with clinically significant abnormalities in laboratory parameters which were deemed clinically significant by the investigator were reported.
Time Frame: Baseline up to Month 14
Population: The safety population was defined as all participants enrolled who had applied study medication at least once.
Measure: Count of Participants; unit: Participants
Groups:
- Adapalene/Benzoyl Peroxide: Participants were treated with Adapalene 0.1 percent % (W/W) and benzoyl peroxide 2.5 % (W/W) gel topically to the face and trunk area, as applicable, once daily in the evening.
Arm/Group | Adapalene/Benzoyl Peroxide
Number analyzed (Participants) | 452
Participants
  Hematology | 0
  Blood Chemistry | 0
  Urine Analysis | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 14 months
Groups:
- Adapalene/Benzoyl Peroxide: Participants were treated with adapalene 0.1 % (W/W) and benzoyl peroxide 2.5 % (W/W) gel topically to the face and truck area, as applicable, once daily in the evening.
Arm/Group | Adapalene/Benzoyl Peroxide
All-Cause Mortality (participants affected / at risk) | 0/452
Serious Adverse Events (participants affected / at risk) | 5/452
Other Adverse Events (participants affected / at risk) | 288/452
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adapalene/Benzoyl Peroxide (N=452)
Major Depression (Psychiatric disorders) | 1
Bipolar Disorder (Psychiatric disorders) | 1
Staphylococcal Infection (Infections and infestations) | 1
Clavicle Fracture (Injury, poisoning and procedural complications) | 1
Syncope (Nervous system disorders) | 1
Drug Abuser (Social circumstances) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adapalene/Benzoyl Peroxide (N=452)
Nasopharyngitis (Infections and infestations) | 30
Upper Respiratory Tract Infection (Infections and infestations) | 26
Influenza (Infections and infestations) | 18
Sinusitis (Infections and infestations) | 15
Pharyngitis Streptococcal (Infections and infestations) | 13
Urinary Tract Infection (Infections and infestations) | 8
Gastroenteritis Viral (Infections and infestations) | 7
Bronchitis (Infections and infestations) | 7
Pharyngitis (Infections and infestations) | 4
Herpes Simplex (Infections and infestations) | 4
Gastroenteritis (Infections and infestations) | 3
Otitis Externa (Infections and infestations) | 3
Labyrinthitis (Infections and infestations) | 3
Otitis Media (Infections and infestations) | 2
Respiratory Tract Infection Viral (Infections and infestations) | 2
Gingival Infection (Infections and infestations) | 2
Ear Infection (Infections and infestations) | 2
Tonsillitis (Infections and infestations) | 2
Vaginal Mycosis (Infections and infestations) | 2
Tinea Pedis (Infections and infestations) | 1
Subcutaneous Abscess (Infections and infestations) | 1
Salmonellosis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Body Tinea (Infections and infestations) | 1
Nail Infection (Infections and infestations) | 1
Tooth Infection (Infections and infestations) | 1
Lower Respiratory Tract Infection (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Helicobacter Gastritis (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Eye Infection (Infections and infestations) | 1
Conjunctivitis Infective (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Abdominal Infection (Infections and infestations) | 1
Upper Respiratory Tract Infection Bacterial (Infections and infestations) | 1
Varicella (Infections and infestations) | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 80
Erythema (Skin and subcutaneous tissue disorders) | 25
Skin Desquamation (Skin and subcutaneous tissue disorders) | 23
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 17
Pruritus (Skin and subcutaneous tissue disorders) | 7
Acne (Skin and subcutaneous tissue disorders) | 5
Swelling Face (Skin and subcutaneous tissue disorders) | 5
Skin Discomfort (Skin and subcutaneous tissue disorders) | 5
Urticaria (Skin and subcutaneous tissue disorders) | 4
Dermatitis Exfoliative (Skin and subcutaneous tissue disorders) | 3
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 3
Dermatitis (Skin and subcutaneous tissue disorders) | 2
Seborrhoeic Dermatitis (Skin and subcutaneous tissue disorders) | 2
Acne Cystic (Skin and subcutaneous tissue disorders) | 2
Rosacea (Skin and subcutaneous tissue disorders) | 1
Dermal Cyst (Skin and subcutaneous tissue disorders) | 1
Pruritus Generalised (Skin and subcutaneous tissue disorders) | 1
Pigmentation Disorder (Skin and subcutaneous tissue disorders) | 1
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 1
Pain of Skin (Skin and subcutaneous tissue disorders) | 1
Heat Rash (Skin and subcutaneous tissue disorders) | 1
Face Odema (Skin and subcutaneous tissue disorders) | 1
Dyshidrosis (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Skin Hypopigmentation (Skin and subcutaneous tissue disorders) | 1
Skin Burning Sensation (Skin and subcutaneous tissue disorders) | 1
Application Site Burning (General disorders) | 64
Application Site Irritation (General disorders) | 18
Pyrexia (General disorders) | 2
Oedema Peripheral (General disorders) | 1
Fatique (General disorders) | 1
Sunburn (Injury, poisoning and procedural complications) | 21
Joint Sprain (Injury, poisoning and procedural complications) | 5
Hand Fracture (Injury, poisoning and procedural complications) | 3
Excoriation (Injury, poisoning and procedural complications) | 3
Arthropod Bite (Injury, poisoning and procedural complications) | 2
Thermal Burn (Injury, poisoning and procedural complications) | 2
Post Procedural Pain (Injury, poisoning and procedural complications) | 2
Tendon Injury (Injury, poisoning and procedural complications) | 2
Muscle Strain (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 1
Skin Laceration (Injury, poisoning and procedural complications) | 1
Chemical Injury (Injury, poisoning and procedural complications) | 1
Joint Dislocation (Injury, poisoning and procedural complications) | 1
Tooth Injury (Injury, poisoning and procedural complications) | 1
Animal Bite (Injury, poisoning and procedural complications) | 1
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Facial Bones Fracture (Injury, poisoning and procedural complications) | 1
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 14
Nasal Conjection (Respiratory, thoracic and mediastinal disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 3
Nasal Odema (Respiratory, thoracic and mediastinal disorders) | 1
Rhitinis (Respiratory, thoracic and mediastinal disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 1
Allergic Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 6
Abdominal Pain Upper (Gastrointestinal disorders) | 4
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 2
Hiatus Hernia (Gastrointestinal disorders) | 2
Gastrointestinal Upset (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastric Ulcer (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Abdominal Pain Lower (Gastrointestinal disorders) | 1
Gingivitis (Gastrointestinal disorders) | 1
Headache (Nervous system disorders) | 21
Migraine (Nervous system disorders) | 2
Convulsion (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 9
Anxiety (Psychiatric disorders) | 4
Attention Deficit/Hyperactivity Disorder (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 2
Drug Dependence (Psychiatric disorders) | 1
Stress Symptoms (Psychiatric disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 6
Tendonitis (Musculoskeletal and connective tissue disorders) | 2
Neck Pain (Musculoskeletal and connective tissue disorders) | 2
Tendon Disorder (Musculoskeletal and connective tissue disorders) | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Laboratory Test Abnormal (Investigations) | 2
Mean Cell Hemoglobin Decreased (Investigations) | 1
Liver Function Test Abnormal (Investigations) | 1
Hepatic Enzyme Increased (Investigations) | 1
Heart Rate Increased (Investigations) | 1
Haemoglobin Increased (Investigations) | 1
Haemoglobin Decreased (Investigations) | 1
Haematocrit Increased (Infections and infestations) | 1
Haematocrit Decreased (Investigations) | 1
Blood Creatinine Increased (Investigations) | 1
Alanine Aminotransferase Increased (Investigations) | 1
White Blood Cell Count Increased (Investigations) | 1
Protein Urine Present (Investigations) | 1
Platelet Count Abnormal (Investigations) | 1
Mean Cell Volume Abnormal (Investigations) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 7
Dysmenorrhoea (Reproductive system and breast disorders) | 4
Amenorrhoea (Reproductive system and breast disorders) | 1
Ovarian Cyst Ruptured (Reproductive system and breast disorders) | 1
Cervical Dysplasia (Reproductive system and breast disorders) | 1
Seasonal Allergy (Immune system disorders) | 3
Food Allergy (Immune system disorders) | 1
Drug Hypersensitivity (Immune system disorders) | 1
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Seborrhoeic Keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dysplastic Naevus Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ear Pain (Ear and labyrinth disorders) | 1
Ear Discomfort (Ear and labyrinth disorders) | 1
Tympanic Membrane Perforation (Ear and labyrinth disorders) | 1
Eyelid Oedema (Eye disorders) | 2
Myopia (Eye disorders) | 1
Eye Discharge (Eye disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Calcus Urinary (Renal and urinary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes